CLINICAL TRIAL: NCT02734771
Title: Phase II Pilot Study of Brentuximab Vedotin, Rituximab and Dose Attenuated CHP in Elderly Patients With DLBCL
Brief Title: A Study of Brentuximab Vedotin, Rituximab, and Dose Attenuated CHP in Elderly Patients With Diffuse Large B-Cell Lymphoma (DLBCL)
Acronym: BV mini CHP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Patrick Reagan (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor-Investigator, Patrick Reagan, Senior Instructor, Hematology/Oncology, University of Rochester
Organization: University of Rochester (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULYM15105; IST-2014-100578 (Other Grant/Funding Number: Seattle Genetics)
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Diffuse Large B-Cell Lymphoma
Keywords: DLBCL
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Brentuximab Vedotin; Rituximab; Cyclophosphamide; Doxorubicin; liposomal doxorubicin; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BV+mini-R-CHP (Experimental): Brentuximab vedotin 1.8 mg/kg IV day 1 for six cycles Rituximab 375 mg/m2 IV day 1 for six cycles Cyclophosphamide 400 mg/m2 IV day 1for six cycles Doxorubicin 25 mg/m2 IV day 1 for six cycles Prednisone 40 mg/m1 PO days 1-5 for six cycles
  Interventions: Drug: Brentuximab vedotin; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone

INTERVENTIONS:
Drug: Brentuximab vedotin
  Other Names: Adcetris; SGN-35; cAC10-vcMMAE
Drug: Rituximab
  Other Names: Rituxan; Mabthera
Drug: Cyclophosphamide
  Other Names: Cytoxan; Lyophilizedcytoxan; Endoxan; Neosar; Procytox; Revimmune; Cycloblastin
Drug: Doxorubicin
  Other Names: Adriamycin; Doxil; Caelyx; Myocet
Drug: Prednisone
  Other Names: Deltasone; Orasone; Adasone; Deltacortisone; Prednisonum

SUMMARY:
This is a study incorporating brentuximab vedotin and dose attenuated rituximab, cyclophosphamide, doxorubicin, and prednisone (R-CHP) into initial therapy for elderly patients with DLBCL. Vincristine will be omitted from the standard R-CHOP regimen given the overlapping toxicities with brentuximab vedotin.

DETAILED DESCRIPTION:
This is a multicenter, single-arm pilot study incorporating brentuximab vedotin and dose attenuated rituximab, cyclophosphamide, doxorubicin, and prednisone (R-CHP) into initial therapy for elderly patients with DLBCL. Vincristine will be omitted from the standard R-CHOP regimen given the overlapping toxicities with brentuximab vedotin. CD30 positivity will be determined at enrollment and patients will be enrolled into a CD30 positive and negative group in equal numbers. Additionally, a Comprehensive Geriatric Assessment (CGA) will be performed on all patients, but this will not be used to guide treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary written informed consent before performance of any study-specific procedure not part of routine medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care. Subjects must be able to understand and be willing to sign the written informed consent form.
* Men and women aged greater than or equal to 75 years of age
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-3
* Histologically-confirmed DLBCL by World Health Organization classification by site hematopathologist

  * Histologic transformation (HT) will be included on the study. This must be confirmed with a biopsy. Patients with HT must not have received an anthracycline-containing regimen in the past.
  * Composite lymphoma containing both indolent and large cell features will be included
* Has received no prior therapy for DLBCL or HT with the exception of a course of prednisone of less than or equal to 7 days given for lymphoma related symptoms; prior therapy for follicular lymphoma is accepted, but no prior anthracycline-containing therapy.
* Carriers of hepatitis B virus should be closely monitored for clinical and laboratory signs of active hepatitis B virus infection and for signs of hepatitis throughout study participation.
* Total bilirubin must be less than 1.5 times the upper limit of normal (ULN) unless the elevation is known to be due to Gilbert syndrome.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) must be less than 3 times the upper limit of the normal range. AST and ALT may be elevated up to 5 times the ULN if their elevation can be reasonably ascribed to the presence of DLBCL in liver.

Exclusion Criteria:

* Patient has a platelet count of ≤50,000/mm3 within 14 days before enrollment.
* Patient has an absolute neutrophil count of < 1,000/mm3 within 14 days before enrollment.
* Patient has a calculated or measured creatinine clearance of <30 mL/minute within 14 days before enrollment.
* Patient is receiving peritoneal dialysis or hemodialysis
* Patient has ≥Grade 2 peripheral neuropathy within 14 days before enrollment.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* New York Heart Association class III heart failure or ejection fraction of less than 30% on echocardiogram or Multi Gated Acquisition Scan (MUGA)
* Patient has received other investigational drugs with 14 days before enrollment
* Prior exposure to anthracycline
* Patient has concomitant active malignancy that the treating physician or PI feels may interfere with the ability to measure the primary or secondary outcomes

  * Patients with a history of curative, surgically treated basal or squamous cell carcinoma or stage 1 melanoma of the skin or in situ carcinoma of the cervix are eligible.
  * Patients with a malignancy that has been treated with surgery alone with curative intent will also be excluded, unless the malignancy has been in documented remission without treatment for ≥ 3 years prior to enrollment.
* Patient is known to be HIV positive (test result not required for enrollment).
* History of solid organ transplantation, or post-transplant lymphoproliferative disorder
* Patient has history of allogeneic stem cell transplantation.
* History of, or clinically apparent central nervous system (CNS) lymphoma
* Any clinically significant abnormality in screening blood chemistry, hematology, or urinalysis results that, in the judgment of the investigator, would impede adequate evaluation of adverse events and/or response to treatment, or that requires aggressive intervention

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-06; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percent of Subjects Completing Regimen | 20 weeks
  Number of subjects who complete all 6 cycles of the therapy divided by the total number of subjects.

SECONDARY OUTCOMES:
Overall Survival | 2 years
  Number of participants who are alive after two years.
Progression Free Survival | 2 years
  Per the Lugano Criteria, progression is defined as an individual node/lesion that increases in size by 50% or in the setting of splenomegaly, the splenic length must increase by 50% of the extent of its prior increase beyond baseline (eg, a 15-cm spleen must increase to 16 cm). If no prior splenomegaly, must increase by at least 2 cm from baseline or any new or recurrent splenomegaly or new or clear progression of preexisting non-measured lesions or regrowth of previously resolved lesions. or assessable disease of any size unequivocally attributable to lymphoma or new or recurrent involvement.
Overall Response Rate | 20 weeks
  The overall response rate is the proportion of subjects who achieve a complete response or partial response based on the Lugano Criteria. Per the Lugano Criteria, complete response is defined as a Deauville score of 1, 2 or 3 and partial response is defined as Deauville score of 4 or 5, but decreased from baseline. Using CT measurements a complete response is defined as decrease in lymph node size to 1.5 cm, while a partial response is a 50% or greater reduction in size in 6 target lesions.
Complete Response Rate | 20 weeks
  Proportion of participants who have a complete response rate. Per the Lugano Criteria, complete response is defined as a Deauville score of 1, 2 or 3 and partial response is defined as Deauville score of 4 or 5, but decreased from baseline. Using CT measurements a complete response is defined as decrease in lymph node size to 1.5 cm, while a partial response is a 50% or greater reduction in size in 6 target lesions.

OTHER OUTCOMES:
Number of participants with impairment in physical function | 20 weeks
  Activities of daily living (ADL): ADLs are measures of self-care. ADL independence will be assessed using the Katz Index of Independence in Activities of Daily Living, commonly referred to as the Katz ADL. The Katz ADL is the most appropriate instrument to assess functional status as a measurement of the client's ability to perform activities of daily living independently. Clinicians typically use the tool to detect problems in performing activities of daily living and to plan care accordingly. The Index ranks adequacy of performance in the six functions of bathing, dressing, toileting, transferring, continence, and feeding. Clients are scored yes/no for independence in each of the six functions. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates impairment.
mean number of falls per participant | 20 weeks
Mean change in objective physical performance | baseline and 20 weeks
  Physical performance will be tested using the short physical performance battery (range 0-12). Impairment is a score of less than or equal to 9.
Mean number of comorbidities | 20 weeks
mean change in mini nutritional assessment | baseline and 20 weeks
  The current MNA® is a 6 question assessment that identifies older adults who are malnourished or at risk of malnutrition. Scale=0-30. A score of less than or equal to 11 indicates impairment.
Number of participants with any documented change in the Older Americans Resources and Services social resources assessment. | baseline and 20 weeks
  This is a descriptive assessment.
mean change in the geriatric depression screen | baseline and 20 weeks
  The Geriatric Depression Scale (GDS) is a 30-item self-report assessment used to identify depression in the elderly. Scale ranges from 0-15 with a score of greater than or equal to 5 signifying impairment.
mean change in cognition score | baseline and 20 weeks
  Cognition will be assessed using the blessed orientation memory-concentration (BOMC) test. The BOMC is a screening tool allowing family members, caregivers, or health care professionals to check for suspected dementia in an elderly. Dementia is described as the progressive loss of memory and at least of one other cognitive area, such as language or behavior. The scale is -20 with a score of greater than 10 signifying impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M Reagan, MD, Principal Investigator — Wilmot Cancer Institute, University of Rochester Medical Center
Locations (2):
- United States (2):
  - James P. Wilmot Cancer Institute, University of Rochester Medical Center, Rochester, New York
  - University of Virginia Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No